CLINICAL TRIAL: NCT02884063
Title: Utilizing Free DNA in Embryo Culture Media for Preimplantation Genetic Screening
Brief Title: Utilizing Free DNA in Embryo Culture for PGT
Status: Completed | Type: Observational
Sponsor: Al Baraka Fertility Hospital (Other)
Collaborators: Ibn Sina Hospital (Other Government); Sadat City University (Other)
Responsible Party: Principal Investigator, Ahmad Mustafa Mohamed Metwalley, IVF laboratory manager, Al Baraka Fertility Hospital
Other Study IDs: NGS-PGT
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Chromosome Abnormalities; Genetic Diseases, Inborn; Mutation
Keywords: PGS; PGD; free embryo DNA; NGS; PGT; PGT-a; PGT-m; PGT-HLA
MeSH Terms: conditions — Chromosome Aberrations; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blastomer for growing IVF embryos culture media with its free DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NGS reading for Media Free DNA: Ability to read the DNA product available in embryo culture media using NGS to have valuable diagnostic image for genetic composition of embryo before implantation.
  Interventions: Procedure: NGS reading for Media Free DNA
- NGS reading for blastomer DNA: DNA extracted from Blastomere used for aneuploidy screening.
  Interventions: Procedure: NGS reading for Media Free DNA

INTERVENTIONS:
Procedure: NGS reading for Media Free DNA — NGS reading for Media Free DNA instead of blstomer biopsy

SUMMARY:
In the way for developing and optimizing protocol to be used as non- invasive methodology used as routine testing for PGS.

This protocol is to be adapted to replace the using of life embryo cells for genetic testing and aneuploidy study as well as for any type of genetic testing including single gene disorder or HLA typing or study.

DETAILED DESCRIPTION:
Compare 100 embryos studied using NGS for chromosomal aneuploidies, and compare the results came from free media DNA with this results.

ELIGIBILITY:
Inclusion Criteria:

* all abnormal/aneuploidy embryos rejected for embryo transfer.

Exclusion Criteria:

* all embryos had unsuccessful diagnosis with blastomere biopsy.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Embryos arranged for PGS study
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
DNA isolation | 2 years
  reading amplified DNA using NGS

SECONDARY OUTCOMES:
NGS evaluation | 2 years
  Free DNA isolation and amplification using WGA
Comparison with cell reading using NGS | 2 years
  compare the obtained result with the results provided collected for the same embryo using its blastomer for PGS

CONTACTS AND LOCATIONS:
Overall Officials: Omima Khamis, PHD, Study Director — Genetic Engineering Institute

IPD SHARING:
Plan to Share IPD: Yes
To publish it when it is completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: once final results released.
Access Criteria: 01-December 2019

REFERENCES:
- See also: Non invasive genetic testing — https://www.deepdyve.com/lp/elsevier/non-invasive-preimplantation-genetic-screening-pgs-free-embryonic-dna-3mDt0ZAPbo